CLINICAL TRIAL: NCT02703324
Title: Pharmacokinetics, Glucodynamics, Safety, and Tolerability of LY900014 in Patients With Type 1 Diabetes Mellitus on Continuous Subcutaneous Insulin Infusion Therapy
Brief Title: A Study of LY900014 Formulation in Participants With Type 1 Diabetes Mellitus Using Insulin Pumps
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 16070; I8B-FW-ITRF (Other: Eli Lilly and Company); 2015-004705-16 (EudraCT Number)
Record Dates: First submitted 2016-03-04; First posted 2016-03-09 (Estimated); Results first posted 2020-04-28 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY900014 (Experimental): LY900014 delivered via an insulin pump as a continuous infusion under the skin with intermittent bolus doses during meals for two 3-day periods
  Interventions: Drug: LY900014
- Insulin Lispro (Active Comparator): Insulin lispro delivered via an insulin pump as a continuous infusion under the skin with intermittent bolus doses during meals for two 3-day periods
  Interventions: Drug: Insulin Lispro

INTERVENTIONS:
Drug: LY900014 — Administered subcutaneously (SC)
  Other Names: Ultra-Rapid Lispro
  Arms: LY900014
Drug: Insulin Lispro — Administered SC
  Arms: Insulin Lispro

SUMMARY:
This study evaluated a blood sugar lowering insulin, LY900014, delivered by an insulin pump continuously under the skin. The study was conducted in participants with type 1 diabetes mellitus to investigate how the human body processed LY900014 and its effect on blood sugar levels when it was delivered via an insulin pump. Side effects and tolerability were be documented.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants with Type 1 Diabetes Mellitus (T1DM) who are receiving insulin therapy via an approved insulin pump
* Have a body mass index (BMI) of 18.5 to 33 kilogram per square meter (kg/m²), inclusive, at screening
* Have blood pressure, pulse rate, electrocardiogram (ECG), blood and urine laboratory test results that are acceptable for the study
* Have had no episodes of severe hypoglycemia in the past 6 months (requiring assistance in treatment by a second party)
* Have venous access sufficient to allow for blood sampling
* Have provided written consent and are willing to follow study procedures and commit to the study duration

Exclusion Criteria:

* Are currently participating in or completed a clinical trial within the last 30 days from a clinical trial or any other type of medical research judged to be incompatible with this study
* Have previously participated or withdrawn from this study
* Have or used to have health problems, laboratory test results, blood pressure or ECG readings that, in the opinion of the doctor, could make it unsafe to participate in the study
* Had blood loss of more than 500 milliliters (mL) within the last month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Neuss, Germany

REFERENCES:
- See also: Click here for more information about this study: A Study of LY900014 in Participants With Type 1 Diabetes Mellitus Using Insulin Pumps — http://www.lillytrialguide.com/EN-US/studies/diabetes/itrf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study compared individualized doses of LY900014 (Test) to insulin lispro (Reference) when delivered via an insulin pump. The study consisted of four, three-day treatment periods, with a maximum of one week between doses in consecutive periods.
Groups:
- Sequence 1, TRTR: T = LY900014 Test. R = Insulin Lispro Reference. In each of four periods, individualized doses of study drug were delivered via an insulin pump as a continuous subcutaneous (SC) infusion with intermittent bolus doses immediately before meals for three days.
- Sequence 2, RTRT; Sequence 3, TTRR; Sequence 4, RRTT; Sequence 5, TRRT; Sequence 6, RTTR: T = LY900014 Test. R = Insulin Lispro Reference. In each of four periods, individualized doses of study drug were delivered via an insulin pump as a continuous SC infusion with intermittent bolus doses immediately before meals for three days.
Period: Period One
Arm/Group | Sequence 1, TRTR | Sequence 2, RTRT | Sequence 3, TTRR | Sequence 4, RRTT | Sequence 5, TRRT | Sequence 6, RTTR
Started | 5 | 5 | 5 | 5 | 5 | 5
Received Study Drug | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period Two
Arm/Group | Sequence 1, TRTR | Sequence 2, RTRT | Sequence 3, TTRR | Sequence 4, RRTT | Sequence 5, TRRT | Sequence 6, RTTR
Started | 5 | 5 | 5 | 5 | 5 | 5
Received Study Drug | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 4 | 5 | 5 | 5
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0
Period: Period Three
Arm/Group | Sequence 1, TRTR | Sequence 2, RTRT | Sequence 3, TTRR | Sequence 4, RRTT | Sequence 5, TRRT | Sequence 6, RTTR
Started | 5 | 5 | 4 | 5 | 5 | 5
Received Study Drug | 5 | 5 | 4 | 5 | 5 | 5
Completed | 5 | 5 (One participant discontinued after Period 3. Did not enter Period 4.) | 4 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period Four
Arm/Group | Sequence 1, TRTR | Sequence 2, RTRT | Sequence 3, TTRR | Sequence 4, RRTT | Sequence 5, TRRT | Sequence 6, RTTR
Started | 5 | 4 (One participant discontinued after Period 3. Did not enter Period 4.) | 4 | 5 | 5 | 5
Received Study Drug | 5 | 4 | 4 | 5 | 5 | 5
Completed | 5 | 4 | 4 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- All Participants: Individualized doses of LY900014 (Test) or insulin lispro (Reference) delivered via an insulin pump as a continuous SC infusion with intermittent bolus doses immediately before meals in four, three-day periods.
Arm/Group | All Participants
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 30

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Insulin Lispro Area Under the Concentration Curve From Time Zero to 5 Hours (AUC[0-5h])
Description: PK: Insulin Lispro AUC(0-5h)
Time Frame: Days 1 and 3: -15, 0, 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, 55, 60, 70, 90, 120, 150, 180, 240, 300 minutes post dose for each treatment
Population: All participants who received both study drugs and had evaluable PK data. For one participant in the Insulin Lispro - Reference group, the insulin lispro PK profile (Period Two, Day 3) was excluded from the mean PK analysis, as there was no absorption phase observed.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: picomole*hour per liter (pmol•h/L)
Groups:
- Insulin Lispro - Reference: Individualized doses of insulin lispro delivered via an insulin pump as a continuous SC infusion with intermittent bolus doses during meals for two 3-day periods.
- LY900014 - Test: Individualized doses of LY900014 delivered via an insulin pump as a continuous SC infusion with intermittent bolus doses during meals for two 3-day periods.
Arm/Group | Insulin Lispro - Reference | LY900014 - Test
Number analyzed (Participants) | 29 | 29
picomole*hour per liter (pmol•h/L)
  Day 1 | 918 (26) | 970 (28)
  Day 3 | 906 (30) | 824 (37)

2. Secondary Outcome: Pharmacodynamics (PD): Area Under the Concentration Curve From Time Zero to 5 Hours (AUC[0-5h]) of Glucose Relative to a Mixed Meal Tolerance Test (MMTT)
Description: PD: AUC(0-5h) of Glucose Relative to a Mixed Meal Tolerance Test (MMTT)
Time Frame: Days 1 and 3: -30, -15, 0, 10, 20, 30, 40, 50, 60, 70, 80, 90, 100, 110, 120, 135, 150, 165, 180, 195, 210, 225, 240, 300 minutes post dose for each treatment
Population: All participants who received study drug and had evaluable PD data.
Measure: Mean (Standard Deviation); unit: milligram*hour/deciliter (mg*h/dL)
Groups:
- Insulin Lispro - Reference: Individualized doses of insulin lispro delivered via an insulin pump as a continuous SC infusion with intermittent bolus doses during meals for two three-day periods.
- LY900014 - Test: Individualized doses of LY900014 delivered via an insulin pump as a continuous SC infusion with intermittent bolus doses during meals for two three-day periods.
Arm/Group | Insulin Lispro - Reference | LY900014 - Test
Number analyzed (Participants) | 29 | 29
milligram*hour/deciliter (mg*h/dL)
  Day 1 | 584 (175) | 567 (172)
  Day 3: number analyzed (Participants) | 28 | 29
  Day 3 | 551 (185) | 628 (210)

ADVERSE EVENTS:
Groups:
- Insulin Lispro - Open Label: Individualized doses of open label insulin lispro delivered via an insulin pump as a continuous SC infusion with intermittent bolus doses between periods.
Arm/Group | Insulin Lispro - Reference | LY900014 - Test | Insulin Lispro - Open Label
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 4/29 | 3/30 | 0/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Lispro - Reference (N=29) | LY900014 - Test (N=30) | Insulin Lispro - Open Label (N=30)
Headache (Nervous system disorders) | 4 (4) | 3 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days